CLINICAL TRIAL: NCT06204679
Title: A Phase 1, Open-Label Study to Assess Comparative Bioavailability and Effect of Food on a Prototype Fixed-Dose Combination of Bemnifosbuvir and Ruzasvir Versus Individual Dosage Forms Taken Concomitantly in Healthy Adult Subjects
Brief Title: Pharmacokinetics of Fixed-Dose Combination Tablet of Bemnifosbuvir and Ruzasvir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AT-01B-005
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — ruzasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FDC Fasting (Experimental): Day 1, Day 7, Day 13
  Interventions: Drug: Bemnifosbuvir (BEM)/Ruzasvir (RZR) FDC under fasting conditions
- FDC Fed (Experimental): Day 1, Day 7, Day 13
  Interventions: Drug: Bemnifosbuvir (BEM)/Ruzasvir (RZR) FDC under fed conditions
- Reference Fasting (Experimental): Day 1, Day 7, Day 13
  Interventions: Drug: Bemnifosbuvir (BEM) and Ruzasvir (RZR) as reference formulation under fasting conditions

INTERVENTIONS:
Drug: Bemnifosbuvir (BEM)/Ruzasvir (RZR) FDC under fasting conditions — A Fixed-Dose Combination of Bemnifosbuvir (BEM) and Ruzasvir (RZR)
  Arms: FDC Fasting
Drug: Bemnifosbuvir (BEM)/Ruzasvir (RZR) FDC under fed conditions — A Fixed-Dose Combination of Bemnifosbuvir (BEM) and Ruzasvir (RZR)
  Arms: FDC Fed
Drug: Bemnifosbuvir (BEM) and Ruzasvir (RZR) as reference formulation under fasting conditions — Bemnifosbuvir (BEM) and Ruzasvir (RZR) as separate formulations
  Arms: Reference Fasting

SUMMARY:
This study will assess comparative bioavailability and effect of food on a prototype fixed-dose combination (FDC) of Bemnifosbuvir (BEM) and Ruzasvir (RZR) in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use two methods of birth control from Screening through 90 days after administration of the last dose of study drug.
* Minimum body weight of 50 kg and body mass index (BMI) of 18-30 kg/m2.
* Willing to comply with the study requirements and to provide written informed consent.

Exclusion Criteria:

* Infected with hepatitis B virus, hepatitis C virus, HIV or SARS-CoV-2.
* Abuse of alcohol or drugs.
* Use of other investigational drugs within 28 days of dosing.
* Concomitant use of prescription medications, or systemic over-the-counter medications.
* Other clinically significant medical conditions or laboratory abnormalities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of FDC compared to reference:(Cmax) | Day 1, Day 7, Day 13
  Maximum plasma concentration (Cmax)
Pharmacokinetics (PK) of FDC compared to reference:(AUC) | Day 1, Day 7, Day 13
  Area under the plasma concentration-time curve (AUC)
Food effect of Fixed Dose Combination of Bemnifosbuvir (BEM)/Ruzasvir (RZR):(Cmax) | Day 1, Day 7, Day 13
  Maximum plasma concentration (Cmax)
Food effect of Fixed Dose Combination of Bemnifosbuvir (BEM)/Ruzasvir (RZR):(AUC) | Day 1, Day 7, Day 13
  Area under the plasma concentration-time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Atea Study Site, Cypress, California, United States